CLINICAL TRIAL: NCT07166848
Title: Pilot Trial of Non-invasive Electrostimulation in Chronic Ocular Graft-vs-Host Disease
Brief Title: Electrostimulation Study for Ocular Graft vs. Host Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhonghui K. Luo, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Zhonghui K. Luo, MD, PhD, Principal Investigator, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025P002105
Record Dates: First submitted 2025-08-20; First posted 2025-09-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Chronic Ocular Graft-versus-host Disease
Keywords: GVHD; Electrostimulation
MeSH Terms: interventions — Electrodes; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The principal investigator and the participants will be masked to treatment. The study staff setting up the device will be the only staff who will know the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrostimulation (Experimental): The experimental group will entail the subject wearing the electrodes on the cheeks and forehead, for 30 minutes WITH amplitude.
  Interventions: Device: Electrodes with Currents
- Sham (Sham Comparator): The placebo group will entail the subject wearing the electrodes on the cheeks and forehead, for 30 minutes WITHOUT amplitude.
  Interventions: Device: Electrodes without Currents

INTERVENTIONS:
Device: Electrodes with Currents — Electrodes will be placed on the cheeks and forehead, and treated with an amplitude of 300 µA for 30 mins
  Other Names: Treatment
  Arms: Electrostimulation
Device: Electrodes without Currents — Electrodes will be placed on the cheeks and forehead, and treated with an no amplitude for 30 mins
  Other Names: Sham
  Arms: Sham

SUMMARY:
This trial is testing to see if electrostimulation treatment (ET) will be effective in treating those with ocular Graft vs. Host Disease.

DETAILED DESCRIPTION:
The trial is to test whether transcutaneous electrical stimulation (TES) may be an effective new type of non-invasive treatment for patients who are diagnosed with chronic ocular Graft-vs-Host Disease. Such a treatment can potentially decrease the need for the patients to apply eye drops frequently, repair the damage caused by chronic ocular Graft-vs-Host Disease, and improve the comfort of the eyes naturally.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic ocular graft vs. host disease (oGVHD) (ICCGVHD criteria probable or definite)
* OSDI score of 22 or higher
* NEI corneal staining score (or modified NEI score) of 2 or higher.

Exclusion Criteria:

* Patients with any open wound on the eyelid.
* Patient with any active cornea ulcer, dacryocystitis, hordeolum, filamentary keratitis, uveitis, retinal detachment, uncontrolled glaucoma or other active pathology per PI's discretion.
* Patient with a pacemaker or ICD.
* Patient currently pregnant or with a potential to be pregnant during the study.
* Patient undergoing any ocular surgical procedure (including intravitreal injections) within the past 3 months.
* Patient undergoing any systemic surgical procedures within 2 months.
* Patient undergoing any non-surgical eyelid procedure such as punctal plugs or punctal cautery within 1 month of study initiation.
* Patients on cytotoxic agents, drugs that inhibit peripheral nerve regeneration (i.e. Gabapentin, Nicotine), radiation therapy, or any other therapy per PI's discretion.
* Patients undergoing immunosuppression regimen change within 1 month of study initiation and/or during the study period.
* Patient who wears contact lens of any kind

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-11-30 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Electrostimulation (ES) Treatment. | 8 Weeks
  To evaluate whether the use of electrostimulation (ES) over a course of 10 treatments (in 8 weeks) will ameliorate symptoms and signs of chronic ocular Graft-vs-Host Disease (oGVHD) and the effect on sub-basal corneal nerve regeneration.

CONTACTS AND LOCATIONS:
Overall Officials: Zhonghui Luo, MD, PhD, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear - Longwood Campus, Boston, Massachusetts, United States